CLINICAL TRIAL: NCT01189981
Title: Effect of Internet, Mobil Applications and SMS-based Encouragements to Intensive Exercise in Adolescents With Congenital Heart Disease
Brief Title: Effect of eHealth Encouragements to Intensive Exercise in Adolescents With Congenital Heart Disease
Acronym: PReVaiL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Susanne Hwiid Klausen, ph.d student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHK 3341; 959515921 (Other: Rigshospitalet)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eHealth intervention (Experimental): Standard lifestyle counseling. Short Message Service (SMS) encouragements for physical activity,
  Interventions: Behavioral: eHealth intervention
- Lifestyle counseling (Active Comparator): Standard lifestyle counseling. No Short Message Service (SMS) encouragements for physical activity.
  Interventions: Behavioral: Lifestyle counseling; Behavioral: eHealth intervention

INTERVENTIONS:
Behavioral: Lifestyle counseling — One health conversation at baseline
  Other Names: Health conversations with chronically ill adolescents
  Arms: Lifestyle counseling
Behavioral: eHealth intervention — SMS based encouragements to intensive exercise
  Other Names: SMS based encouragements to intensive exercise

SUMMARY:
All over the world 0.8 % of all live children are born with a Congenital Heart Disease (CHD) due to genetic end environmental causes. Advanced treatment and care has enhanced survival substantially, and adults with CHD are a growing population requiring continuous monitoring and care. Presently 25% of young adults acquire complicating Cardio Vascular Diseases (CVD) in young adulthood amongst other co-morbidities.

It is known that adolescents with CHD are not as physical fit (PF) as their cardiac capability allows, most likely for reasons concerning safety, ability plus inactive everyday life. However, in 2006 The European Society of Cardiology states, that regular exercise at recommended levels can be performed and should be encouraged in all patients with CHD. Training programmes in hospitals have an effect on PF and Quality of Life (QoL) for the few, as most adolescents' find it impossible to fit into everyday life.

It is the investigators hypothesis that an eHealth intervention, to facilitate intensive exercise in the patients' neighbourhood environs, may improve physical fitness more efficiently than standard lifestyle education.

The purpose of the study is to create evidence to recommend an efficient, fun and safe cardiac rehabilitation programme to adolescents with CHD.

Primary outcome measure

Cardiopulmonary exercise capacity: Online V02 max bicycle test

Secondary outcome measure

Level of physical exercise: Actigraph and Questionnaire

Tertiary outcome measure

Quality of Life: PedsQl

Prevail is a national prospective, randomized clinical trial including 216 adolescents aged 13-16 years, who have had cardiac surgery in childhood owing to complex CHD. The patients included are all recommended to be as physical active as their healthy peers and pursue the principle guideline from The National Board of Health: "All children and young people must be physically active for at least 60 minutes a day, preferably longer". Patients with mental retardation and FEV1 at baseline < 80% of predicted are excluded.

The risk of participating in the purposed trial is not regarded as higher than everyday daily living.

Results will be interpreted according to affiliation to health related fitness clusters.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease with allowance for unrestricted exercise
* Diagnosis: Q20.0 Truncus arteriosus communis, Q20.1 Transpositio vasorum incompleta, Q20.3 Transpositio vasorum completa, Q20.5 Inversio ventriculorum cordis, Q21.2 Defectus septi atrioventriculorum cordis, Q21.3 Tetralogia Steno-Fallot, Q22.4 Tricusspidalatresia , Q22.5 Anomalia Ebstein, Q23.2 Mitralatresia, Double outlet right ventricle, Q23.3 Hypoplasia ventriculi sinistri cordis syndrome, Q23.3 Hypoplasia ventriculi dextrii cordis syndrome, Q24.4 Stenosis subaortae congenita, Q25.1 Coarctatio aortae, Q25.1 Coarctatio Aortae, Double inlet left ventricle, Q25.3 Stenosis aortae supravalvularis, Q25.5 Pulmonalatresia.
* Successful Total Cavo Pulmonal Connex (TCPC procedure)
* 13- 16 years of age

Exclusion Criteria:

* Mental retardation
* Untreated asthma
* Syndromes related to CHD

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary exercise capacity | 12 months
  Online V02 max bicycle test

SECONDARY OUTCOMES:
Level of physical exercise | 12 months
  Actigraph and Questionnaire
Quality of Life | 12 months
  PedsQl

CONTACTS AND LOCATIONS:
Overall Officials: Lars Søndergaard, MD, DMSc, Study Director — Rigshospitalet, Denmark; Susanne Klausen, MSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University Hospital Copenhagen, Copenhagen, RegionH, Denmark

REFERENCES:
- [Derived] Klausen SH, Andersen LL, Sondergaard L, Jakobsen JC, Zoffmann V, Dideriksen K, Kruse A, Mikkelsen UR, Wetterslev J. Effects of eHealth physical activity encouragement in adolescents with complex congenital heart disease: The PReVaiL randomized clinical trial. Int J Cardiol. 2016 Oct 15;221:1100-6. doi: 10.1016/j.ijcard.2016.07.092. Epub 2016 Jul 16. PMID 27448540
- See also: A detailed statistical analysis plan for the results of the PReVaiL trial — http://www.rigshospitalet.dk/menu/AFDELINGER/Juliane+Marie+Centret/Forskning/ForskningsenhedenKBS/Forskning/Forskningsmedarbejdere/Susanne+Hwiid+Klausen.htm